CLINICAL TRIAL: NCT06782646
Title: Assessing the Sex-specific, Lipid- and Lipoprotein-lowering Effects of Berberine Using Randomized, Placebo-controlled, Double-masked Trial
Brief Title: Study on the Sex-specific, Lipid- and Lipoprotein-lowering Effects of Berberine
Status: Enrolling by invitation | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Jie Zhao, Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 21222191
Record Dates: First submitted 2025-01-10; First posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Hyperlipidemia
Keywords: Hyperlipidemia; berberine; lipoprotein; lipid; sex-hormones; apoA1; apoB; Lp(a)
MeSH Terms: conditions — Hyperlipidemias | interventions — Berberine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Berberine Group (Experimental): berberine (500 mg orally twice a day)
  Interventions: Drug: Berberine
- Placebo Group (Placebo Comparator): placebo (500 mg orally twice a day)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Berberine — Participants will take purified berberine (500 mg orally twice a day) for 12 weeks.
  Other Names: Berberine (500 mg orally twice a day)
  Arms: Berberine Group
Drug: Placebo — Participants will take placebo tablets, a look-alike substance that contains no drug, (500 mg orally twice a day) for 12 weeks.
  Other Names: Placebo (500 mg orally twice a day)
  Arms: Placebo Group

SUMMARY:
The goal of this clinical trial is to learn if berberine works to affect lipids and lipoproteins in Chinese females aged 20 to 65 years with hyperlipidaemia. The goal also includes to examine the sex-specific effect of berberine on lipids and lipoproteins. Our previous HMRF-funded randomized trial in men and prior evidence suggests berberine affects sex hormones. Given the different sex hormone profiles in men and women, the main question it aims to answer is:

• Does berberine have sex-specific lipid-modifying effects? Researchers will compare berberine to a placebo (a look-alike substance that contains no drug) to see if berberine works to affect lipids and lipoproteins.

Participants will:

* Take a baseline questionnaire
* Take berberine or a placebo every day for 12 weeks
* Take follow-up visits after 8 weeks and 12 weeks for blood sample collections and tests

DETAILED DESCRIPTION:
The overall aim of the project is to assess the sex-specific effects of berberine on lipids, apoA1, apoB, and Lp(a). Specifically, the objectives of the project are to 1) assess the effect of berberine on lipids (total cholesterol, LDL-cholesterol, HDL-cholesterol, non-HDL cholesterol, and TG), lipoproteins (apoA1, apoB, and Lp(a)) and sex hormones by conducting a randomized, parallel, double-masked, placebo-controlled trial of berberine RCT in women; 2) assess the effect of berberine on apoA1, apoB, Lp(a) and sex hormone binding globulin (SHBG) in men using stored samples from our completed RCT of berberine in men; 3) assess whether the effects of berberine on lipids, lipoproteins and sex hormones differ in men and women.

This is a randomized, parallel, double-blinded, placebo-controlled trial of berberine in 100 Chinese women with hyperlipidemia in Hong Kong.

Participants will be randomized to two arms in which half of the participants will receive berberine (500 mg orally twice a day) and the other half will receive placebos (500 mg orally twice a day) for 12 weeks. Blood samples will be taken at baseline, 8-week and 12-week intervention.

The investigators will use an intention-to-treat analysis. Changes in lipids and lipoproteins after 8- and 12-week treatment will be assessed using analysis of variance and generalized estimating equation (GEE) model accounting for measurements at both time points.

ELIGIBILITY:
Inclusion Criteria:

* Women, who are:

  1. aged 20 to 65 years.
  2. of Chinese ethnicity.
  3. with hyperlipidemia, defined as TG greater than 150 mg/dl (1.70 mmol/L), total cholesterol greater than 200 mg/dl (5.16 mmol/L), and/or LDL-cholesterol greater than 100 mg/dl (2.58 mmol/L).
  4. willing to make return visits.
  5. not currently receiving hormone replacement therapy or medications/pills containing hormones (such as hormonal contraception or hormone replacement therapy) in the past 12 months.
  6. not currently taking berberine or nutraceuticals that contain berberine.
  7. free of any congenital diseases, including familial hypercholesterolemia.
  8. free of Glucose-6-Phosphate Dehydrogenase (G6PD) deficiency. G6PD will be tested using G6PD rapid diagnostic tests.
  9. free of hemolytic anemia.
  10. free of any infectious diseases, e.g., seasonal influenza.
  11. without liver/renal diseases.
  12. not pregnant or planning to get pregnant in the next three months. Pregnancy will be ruled out using HCG ULTRA pregnancy tests.
  13. not currently breastfeeding.

Exclusion Criteria:

* All men, and women who did not meet the aforementioned inclusion criteria and/or were unable or unwilling to provide consent.

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Total cholesterol in mmol/L | 4 months for biomarker assessment, 6 months for data analysis
  Total cholesterol, LDL-cholesterol, TG, apoB, and Lp(a), which are causal factors for coronary heart disease.
LDL-cholesterol in mmol/L | 4 months for biomarker assessment, 6 months for data analysis
  Total cholesterol, LDL-cholesterol, TG, apoB, and Lp(a), which are causal factors for coronary heart disease.
Triglycerides in mmol/L | 4 months for biomarker assessment, 6 months for data analysis
  Total cholesterol, LDL-cholesterol, TG, apoB, and Lp(a), which are causal factors for coronary heart disease.
Apolipoprotein B in mg/dL | 4 months for biomarker assessment, 6 months for data analysis
  Total cholesterol, LDL-cholesterol, TG, apoB, and Lp(a), which are causal factors for coronary heart disease.
Lipoprotein (a) in mg/dL | 4 months for biomarker assessment, 6 months for data analysis
  Total cholesterol, LDL-cholesterol, TG, apoB, and Lp(a), which are causal factors for coronary heart disease.

SECONDARY OUTCOMES:
HDL-cholesterol in mmol/L | 4 months for biomarker assessment, 6 months for data analysis
  Other relevant lipids and lipoproteins.
Non-HDL-cholesterol in mmol/L | 4 months for biomarker assessment, 6 months for data analysis
  Other relevant lipids and lipoproteins.as liver and kidney function.
Apolipoprotein A1 in mg/dL | 4 months for biomarker assessment, 6 months for data analysis
  Other relevant lipids and lipoproteins.
Estradiol (E2) in pg/mL | 4 months for biomarker assessment, 6 months for data analysis
  Examine the sex-specific effects of berberine on apoA1, apoB, Lp(a) and lipids
Sex hormone binding globulin (SHBG) in nmol/L | 4 months for biomarker assessment, 6 months for data analysis
  Examine the sex-specific effects of berberine on apoA1, apoB, Lp(a) and lipids
Testosterone in ng/dL | 4 months for biomarker assessment, 6 months for data analysis
  Examine the sex-specific effects of berberine on apoA1, apoB, Lp(a) and lipids

CONTACTS AND LOCATIONS:
Overall Officials: Jie Zhao, Dr, Principal Investigator — The University of Hong Kong
Locations (1):
- School of Public Health, The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided